CLINICAL TRIAL: NCT02451553
Title: Phase I/IB Multi-center Study of Irreversible EGFR/HER2 Tyrosine Kinase Inhibitor Afatinib (BIBW 2992) in Combination With Capecitabine for Advanced Solid Tumors and Pancretico-Biliary Cancers
Brief Title: Afatinib Dimaleate and Capecitabine in Treating Patients With Advanced Refractory Solid Tumors, Pancreatic Cancer or Biliary Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9078; NCI-2015-00684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9078 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1715055 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-05-19; First posted 2015-05-22 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Advanced Malignant Solid Neoplasm; Bile Duct Carcinoma; Recurrent Malignant Solid Neoplasm; Recurrent Pancreatic Carcinoma; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IVA Pancreatic Cancer; Stage IVB Pancreatic Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms | interventions — Afatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (afatinib dimaleate, capecitabine) (Experimental): Patients receive afatinib dimaleate PO QD on days 1-21 and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib Dimaleate; Drug: Capecitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Afatinib Dimaleate — Given PO
  Other Names: (2E)-N-(4-((3-Chloro-4-fluorophenyl)amino)-7-(((3S)-tetrahydrofuran-3-yl)oxy)quinazolin- 6-yl)-4-(dimethylamino)but-2-enamide bis(hydrogen (2Z)-but-2-enedioate); BIBW 2992MA2; BIBW2992 MA2; Gilotrif
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of afatinib dimaleate when given together with capecitabine in treating patients with solid tumors, pancreatic cancer, or biliary cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment and has not responded to previous treatment. Afatinib dimaleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving afatinib dimaleate together with capecitabine may be a better treatment for solid tumors, pancreatic cancer, or biliary cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety, maximum tolerated dose (MTD), and the recommended phase II dose (RP2D) of afatinib dimaleate (afatinib) in combination with capecitabine in patients with advanced solid tumors (phase I) and pancreatico-biliary cancers (phase Ib). (Phase I/Ib)

SECONDARY OBJECTIVES:

I. Evaluate biomarkers of response from tumor biopsies, including markers related to the epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER2) pathways via OncoPlex or other equivalent gene sequencing assay. (Phase I/Ib)

II. Evaluate rates of response and stable disease, duration of response, time to progression, progression-free and overall survival. (Phase I/Ib)

OUTLINE: This is a phase I, dose-escalation study of afatinib dimaleate followed by a phase Ib study.

Patients receive afatinib dimaleate orally (PO) once daily (QD) on days 1-21 and capecitabine PO twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

PHASE I:

* PHASE I: Histologically confirmed solid tumor malignancy
* PHASE I: Life expectancy >= 12 weeks
* PHASE I: No limit on the number of prior systemic therapies for metastatic disease
* PHASE I: Prior treatment with erlotinib, gefitinib or EGFR-blocking monoclonal antibodies (cetuximab and panitumumab) is allowed
* PHASE I: Signed informed consent
* PHASE I: Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* PHASE I: Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* PHASE I: Must be willing to provide tumor tissue biopsy samples (may be fresh or archival paraffin embedded) at baseline
* PHASE I: In order to perform a retrospective biomarker analysis with the next generation gene sequencing UW-OncoPlex assay; fresh tumor biopsies from metastatic or primary tumor lesion will be done if considered safe and feasible by treating physician and radiologist; Patients who already have OncoPlex or other equivalent gene sequencing assay (eg Foundation One, Perthera, Caris etc) test results available from prior tumor biopsy are eligible to participate, without the needed of a repeat tumor biopsy, but the test results need to be provided to the study principal investigator
* PHASE I: Females of childbearing potential must use an effective method of contraception (barrier method of birth control or abstinence) from the time of consent until at least 180 days following discontinuation of protocol therapy; females of childbearing potential must have a negative pregnancy test within 3 days prior to registration for protocol therapy; patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months; females must not be pregnant or breastfeeding; in rare cases of an endocrine-secreting tumor, human chorionic gonadotropin (hCG) levels may be above normal limits (falsely-positive) but with no pregnancy in the patient; in these cases, there should be a repeat serum hCG test (with a non-rising result) to rule out pregnancy; upon confirmation of results and discussion with the Sponsor-Investigator, these patients may enter the study
* PHASE I: Sexually active male subjects must use an effective method of contraception (barrier method of birth control or abstinence) from the time of consent until at least 180 days following discontinuation of protocol therapy
* PHASE I: Absolute neutrophil count >= 1500/uL
* PHASE I: Platelet count >= 100,000/uL
* PHASE I: Hemoglobin >= 9 gm/dL
* PHASE I: Total bilirubin =< 1.5 times upper limit of normal (ULN)
* PHASE I: Transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) =< 2.5 x ULN
* PHASE I: Prothrombin time (PT) (or international normalized ratio [INR]) and partial thromboplastin time (PTT) =< 1.5 x ULN
* PHASE I: Calculated creatinine clearance (CrCl) >= 60 mL/min calculated by Cockcroft-Gault formula

PHASE IB:

* PHASE IB: Histologically confirmed refractory locally-advanced unresectable or metastatic pancreatic or biliary cancer
* PHASE IB: Life expectancy >= 12 weeks
* PHASE IB: =< 2 lines of prior systemic therapy for metastatic disease (if patients have metastatic disease)
* PHASE IB: =< 2 lines of prior systemic therapy for patients with progressive locally-advanced disease
* PHASE IB: No prior treatment with erlotinib is allowed for pancreatic cancer patients
* PHASE IB: ECOG PS 0-1
* PHASE IB: Signed informed consent
* PHASE IB: Measurable disease according to RECIST v1.1
* PHASE IB: Must be willing to provide tumor tissue biopsy samples (may be fresh or archival paraffin embedded) at baseline
* PHASE IB: Fresh tumor biopsies from metastatic or primary tumor lesions will be done only if considered safe and feasible by treating physician and radiologist; patients who already have OncoPlex or other equivalent gene sequencing assay (eg Foundation One, Perthera, Caris etc) test results available from prior tumor biopsy are eligible to participate, without the needed of a repeat tumor biopsy, but the test results need to be available to the study principal investigator
* PHASE IB: Females of childbearing potential must use an effective method of contraception (barrier method of birth control or abstinence) from the time of consent until at least 180 days following discontinuation of protocol therapy; females of childbearing potential must have a negative pregnancy test within 3 days prior to registration for protocol therapy; patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months; females must not be pregnant or breastfeeding; in rare cases of an endocrine-secreting tumor, hCG levels may be above normal limits (falsely-positive) but with no pregnancy in the patient; in these cases, there should be a repeat serum hCG test (with a non-rising result) to rule out pregnancy; upon confirmation of results and discussion with the sponsor-investigator, these patients may enter the study
* PHASE IB: Sexually active male subjects must use an effective method of contraception (barrier method of birth control or abstinence) from the time of consent until at least 180 days following discontinuation of protocol therapy
* PHASE IB: Patients in the expansion cohort must have a measurable site of disease according to RECIST (v 1.1) that has not been previously irradiated, or evidence of at least 20% progression in a previously irradiated lesion, and assessed by imaging within 28 days prior to registration for protocol therapy
* PHASE IB: Absolute neutrophil count >= 1500/uL
* PHASE IB: Platelet count >= 100,000/uL
* PHASE IB: Hemoglobin >= 9 gm/dL
* PHASE IB: Total bilirubin =< 1.5 times upper limit of normal (ULN)
* PHASE IB: Transaminases (AST and/or ALT) =< 2.5 x ULN
* PHASE IB: PT (or INR) and PTT =< 1.5 x ULN
* PHASE IB: Calculated creatinine clearance (CrCl) >= 60 mL/min calculated by Cockcroft-Gault formula

Exclusion Criteria:

* Prior treatment with afatinib
* Untreated or symptomatic brain metastases requiring corticosteroid therapy (no corticosteroid use for this purpose in the preceding 4 weeks)
* Diagnosis with any of the following in the 12 months prior to registration: severe/unstable angina, myocardial infarction, uncontrolled cardiac arrhythmia, congestive heart failure, cerebrovascular accident or transient ischemic attack
* Active venous thrombosis with contraindication for anticoagulation
* Patients taking warfarin; if anticoagulation is required, the patient must be on a stable dose of a Food and Drug Administration (FDA) approved anticoagulant other than warfarin (e.g. enoxaparin, dalteparin, fondaparinux, apixaban, rivaroxaban) for at least 30 days
* Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient?s ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
* Gastrointestinal tract disease or any other reasons resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, active peptic ulcer disease or chronic diarrhea
* History of bone marrow transplant and stem cell rescue
* Receipt of any chemotherapy, biological therapy or investigational agents within 3 weeks prior to study registration
* Radiotherapy within 4 weeks prior to therapy except palliative radiation to target organs other than primary tumor may be allowed up to 2 weeks prior to registration
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Known pre-existing interstitial lung disease
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn?s disease, ulcerative colitis, chronic diarrhea, malabsorption)
* Known active hepatitis B infection (defined as presence of hepatitis B [HepB] surface antigen [sAg] and/or Hep B deoxyribonucleic acid [DNA]), known active hepatitis C infection (defined as presence of hepatitis C [Hep C] ribonucleic acid [RNA]) and/or known human immunodeficiency virus (HIV) carrier

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days following the last dose of study treatment
  Adverse events will be tabulated and summarized by dose levels. Summary tabulations will be presented displaying the number of observations, mean, standard deviation, median, minimum, and maximum for continuous variables, and the number and percentage per category for categorical data. Toxicity measurement will be accompanied by 90% confidence intervals.
Incidence of dose limiting toxicity (DLT) graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase Ib) | Up to 21 days
  DLTs will be tabulated and summarized by dose levels. Summary tabulations will be presented displaying the number of observations, mean, standard deviation, median, minimum, and maximum for continuous variables, and the number and percentage per category for categorical data. Toxicity measurement will be accompanied by 90% confidence intervals.
Maximum tolerated dose (MTD) of afatinib dimaleate in combination with capecitabine (Phase Ib) | Up to 21 days
  Defined as the dose at which 0/3 or =< 1/6 patients experience a DLT graded according to NCI CTCAE version 4.0, will be assessed.
Recommended phase 2 dose (RP2D) (Phase Ib) | Up to 3 years
  Defined as the best tolerated dose overall, considering overall toxicity, including beyond course 1, will be evaluated.

SECONDARY OUTCOMES:
Biomarker profile (including EGFR and HER2 gene copy number and mutations, Kirsten rat sarcoma viral oncogene homolog, B-Raf proto-oncogene, serine/threonine kinase, neuroblastoma RAS viral oncogene homolog NRAS mutations, and E-cadherin expression) | Baseline
  Will be summarized using mean +/- standard deviation. Baseline biomarker profile will also be summarized by the categories of treatment responses. Logistic models with objective response and stable disease as outcome and the baseline tumor profile as covariate will be fitted to evaluate their association. Correlative analysis of the presence of specific biomarkers and objective response/stable disease and progression free survival (PFS) (for patients in expansion cohorts) will be performed using Chi-square test or Fisher?s exact tests, as appropriate.
Duration of response | Time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
  Duration of response will be assessed with the Kaplan-Meier method.
Duration of stable disease | Time that stable disease is documented until the first date that recurrent disease is objectively documented, assessed up to 3 years
  Duration of stable disease will be assessed with the Kaplan-Meier method.
Overall survival | From the day of first treatment to the earlier of (1) death (from any cause) and (2) the last date of subject contact, assessed up to 3 years
  Overall survival will be assessed with the Kaplan-Meier method.
Progression-free survival | From time from registration to disease progression or death of any cause, assessed up to 3 years
  Assessed with the Kaplan-Meier method.
Rates of response, assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 3 years
  Response rates will be tabulated and summarized by dose levels. Response rate measurement will be accompanied by 90% confidence intervals.
Stable disease, defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to quality for progressive disease assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 3 years
  Stable disease will be tabulated and summarized by dose levels.
Time to progression | From the study enrollment until the criteria for disease progression are met (or death occurs), assessed up to 3 years
  Time to progression will be assessed with the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Elena G. Chiorean, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No